CLINICAL TRIAL: NCT00806507
Title: Early Detection and Prediction of Chemotherapy Induced Cardiac Toxicity in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0339
Record Dates: First submitted 2008-11-20; First posted 2008-12-10 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: Tissue Doppler Imaging; B-type natriuretic peptide; Advia Centaur immunoassay system; GE Vivid ultrasound machine; Roche 2010 system; Echocardiography; Herceptin
MeSH Terms: conditions — Breast Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Echocardiogram + Blood Test: Additional Echocardiogram views performed in 5-10 minutes of regularly scheduled echocardiograms plus blood tests measuring of hormones and metabolic proteins (such as sugars and acids).
  Interventions: Procedure: Echocardiograms; Procedure: Blood Test

INTERVENTIONS:
Procedure: Echocardiograms — Additional views performed in 5-10 minutes of regularly scheduled echocardiograms.
Procedure: Blood Test — Measuring of hormones and metabolic proteins (such as sugars and acids).

SUMMARY:
The goal of this clinical research study is to learn whether different ways of viewing echocardiogram pictures along with blood tests can help to see heart-related side effects of chemotherapy and trastuzumab earlier than the usual tests.

DETAILED DESCRIPTION:
Echocardiogram:

Because of the heart-related side effects of chemotherapy and trastuzumab, your regular doctor will monitor your heart's function as part of your routine care. You will have echocardiograms performed before you begin treatment, and then every 3 months. An echocardiogram uses sound waves to check your heart's health.

If you decide to take part in this study, researchers will take several additional pictures of your heart during each of your regularly scheduled echocardiograms. The additional pictures will make the procedure take about 5-10 minutes longer than the regular echocardiogram. These pictures will be viewed in a different way than the standard echocardiogram pictures. Researchers hope viewing the pictures this way can help researchers to find heart problems earlier than the usual tests.

Blood Tests:

Blood (about 4 teaspoon each time) will be drawn during the routine blood draw that occurs closest to the regularly scheduled echocardiograms.

The heart produces hormones called BNP and NT-proBNP. These hormones can be measured in the blood. BNP and NT-proBNP levels can be higher when the heart is not working as well. Researchers will measure these hormones at the time of each echocardiogram. Researchers hope to learn whether measuring these hormones can help identify the heart-related side effects of chemotherapy and trastuzumab earlier than the usual tests.

Researchers will also measure metabolic proteins (such as sugars and acids) in the blood. Researchers hope to learn whether measuring these metabolic proteins can help identify the heart-related side effects of chemotherapy and trastuzumab earlier than the usual tests.

Because protein, sugar or acid levels may be temporarily changed after you eat, you will be asked not to eat overnight before having your blood drawn.

Study Visits:

You will have 6 study visits around the time that you have an echocardiogram. These visits will occur before you take Herceptin, when you begin Herceptin, and 3, 6, 9, and 12 months later. These study visits will be scheduled on days when you are already making a visit to your regular doctor. You will not have to make any special visits to the hospital for this research study.

During each study visit, you will be asked about any symptoms you may be experiencing, and any medications you may be taking. Your blood pressure and heart rate will be measured.

You will also take a quality of life questionnaire at each study visit. This questionnaire asks you how the cancer may have interfered with your daily life. It should take about 15 minutes to complete.

Length of Study:

You will be considered off-study once you complete the 6 study visits.

This is an investigational study. Up to 100 patients will take part in this multicenter study. Up to 20 patients will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. HER-2 positive breast cancer
3. Scheduled to receive Herceptin infusion therapy after exposure to anthracycline-based chemotherapy in one of the following manners: Adjuvant or neoadjuvant treatment with anthracycline-based chemotherapy preceded or followed by Herceptin infusion therapy, Herceptin monotherapy in patients with metastatic disease previously treated with anthracycline-based chemotherapy, Herceptin in combination with non-anthracycline chemotherapy in patients with metastatic disease previously treated with anthracycline-based chemotherapy
4. Normal baseline left ventricular ejection fraction.

Exclusion Criteria:

1. Pre-existing cardiomyopathy (Left Ventricular Ejection Fraction (LVEF) < 50%)
2. Other contraindication to Herceptin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients treated with chemotherapy and Herceptin (trastuzumab)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2008-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Predictors of cardio-toxicity in female patients with breast cancer exposed to trastuzumab +/- previous anthracycline agents | Baseline to 12 months
  Identification of heart-related side effects of chemotherapy and trastuzumab using echocardiogram pictures plus blood tests.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Banchs, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Partners Healthcare Systems, Boston, Massachusetts
  - UT MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org